CLINICAL TRIAL: NCT06938204
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Multiple Ascending Dose, and Food-Effect Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetics of INV-101 Administered Orally to Healthy Adult Subjects
Brief Title: Single Ascending Dose, Multiple Ascending Dose, Food Effect Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: INV101-02
Record Dates: First submitted 2025-04-03; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Intervention Model Description: 8 subjects were randomized to 6 Active and 2 Placebo in each cohort.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- SAD A (Experimental)
  Interventions: Drug: INV-101; Drug: INV-101 Placebo
- SAD B (Experimental)
  Interventions: Drug: INV-101; Drug: INV-101 Placebo
- SAD C (Experimental)
  Interventions: Drug: INV-101; Drug: INV-101 Placebo
- MAD A (Experimental)
  Interventions: Drug: INV-101; Drug: INV-101 Placebo
- MAD B (Experimental)
  Interventions: Drug: INV-101; Drug: INV-101 Placebo
- MAD C (Experimental)
  Interventions: Drug: INV-101; Drug: INV-101 Placebo

INTERVENTIONS:
Drug: INV-101 — SAD MAD
Drug: INV-101 Placebo — SAD MAD

SUMMARY:
This is a 2-part study. Parts 1 and 2 will be a randomized, double-blind, placebo-controlled investigations of SAD (Part 1) and MAD (Part 2) of orally administered INV-101 in healthy adult subjects. Food effect will also be assessed in one cohort in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects must follow protocol specified contraception guidance as described in Section 7.4.5 and agree to refrain from sperm donation until 90 days after the last dosing.
* Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing based on subject self-reporting.
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at the screening visit.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, or vital signs, as deemed by the PI or designee at the screening visit, including the following:

Exclusion Criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing.
5. History or presence of hypersensitivity or idiosyncratic reaction to compounds related to the study drug or study drug excipients.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Safety Analysis | 7 days after last dosing
  Adverse Events:
  AEs will be coded using the most current version of Medical Dictionary for Regulatory Activities® (MedDRA®). A by-subject AE data listing, including verbatim term, preferred term, treatment (INV-101 or placebo), severity, and relationship to drug, will be provided. The number of subjects experiencing treatment-emergent adverse events (TEAEs) and the number of TEAEs will be summarized by study part and treatment (INV-101 or placebo) using frequency counts.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 3 days
  AUC0-12, AUC0-t, AUC0-inf
Peak Plasma Concentration (Cmax) | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No